CLINICAL TRIAL: NCT07100704
Title: A Phase II Clinical Trial Evaluating the Efficacy and Safety of Nivolumab Monotherapy for Incurable Recurrent or Metastatic Olfactory Neuroblastoma.
Brief Title: Recurrent/Metastatic Olfactory Neuroblastoma: Evaluating the Efficacy and Safety of Nivolumab
Acronym: Orion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Japan Research Foundation for Clinical Pharmacology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Orion; jRCT1031240654 (Other: Ministry of Health, Labour and Welfare)
Record Dates: First submitted 2025-07-10; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Recurrent/ Metastatic Olfactory Neuroblastoma
Keywords: Recurrent/ Metastatic Olfactory Neuroblastoma; Nivolumab
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The decision on which treatment to administer will be made through consultation between the participant in this trial and their attending physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab monotherapy (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 240 mg will be administered on Day 1 and Day 15 of each cycle, or 480 mg will be administered on Day 1 of each cycle, and this will be continued until disease progression. One cycle is 28 days. The decision on which treatment to administer will be made through consultation between the participant in this trial and the site principal investigator or site co-investigator.

SUMMARY:
This trial evaluates the efficacy and safety of nivolumab monotherapy in patients with recurrent or metastatic olfactory neuroblastoma that is difficult to treat with curative intent. Specifically, nivolumab 240 mg will be administered on Day 1 and Day 15 of each cycle, or nivolumab 480 mg will be administered on Day 1 of each cycle, and this will be continued until disease progression. One cycle is 28 days. The decision on which treatment to administer will be made through consultation between the participant in this trial and their attending physician.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Age ≥ 18 years.
3. Histologically confirmed olfactory neuroblastoma.
4. Not eligible for curative local therapy (surgery/radiation).
5. Histological confirmation from recurrent/metastatic lesion or PET-CT evidence.
6. Disease progression after prior chemotherapy.
7. ECOG Performance Status 0-1.
8. Expected survival ≥ 3 months.
9. At least one measurable lesion per RECIST v1.1.
10. Adequate organ function; (1) Absolute Neutrophil Count ≥ 1,000/mm³ (2) Hemoglobin ≥ 8.0 g/dL (3) Platelets ≥ 75,000/mm³ (4) Total bilirubin ≤ 1.5×ULN (≤3.0×ULN for constitutional hyperbilirubinemia) (5) AST/ALT ≤ 3×ULN (≤5×ULN with liver metastasis) (6) Serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 40 mL/min
11. If the participant is female, she agrees to use contraception and refrain from breastfeeding during the treatment and for 5 months after the treatment. If the participant is male, he agrees to use contraception during the treatment and for 7 months after the treatment.

Exclusion Criteria:

1. Active progressive multiple primary cancers (synchronous multiple cancers and metachronous multiple cancers with a disease-free interval of 5 years or less. However, lesions equivalent to carcinoma in situ or mucosal cancer that are considered curable by local treatment are not included as multiple primary cancers. Additionally, this may not apply if the attending physician determines that early-stage cancer will not be a prognostic factor.).
2. Has a systemic infection that requires treatment.
3. It has been determined that one is infected with HIV or AIDS-related diseases.
4. Having an active autoimmune disease that required systemic therapy.
5. Having interstitial lung disease.
6. Pregnant or breastfeeding.
7. Any other cases where the attending physician determines that the treatment in this protocol is inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-04-14 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Through study completion, assessed up to 3 years.
  Based on the judgment by the Investigator or Sub-investigator, according to the Response evaluation criteria in solid tumors (RECIST) guideline version 1.1. The proportion of participants who complete response (CR) or partial response (PR) will be confirmed for overall response according to RECIST version 1.1.

SECONDARY OUTCOMES:
Duration of Response | Through study completion, assessed up to 3 years.
  The period from when CR or PR was first confirmed in the overall effect, according to the RECIST version. 1.1, to the earlier date when progression (PD based on imaging diagnosis) was determined or the date of death due to any cause.
Best Overall Response | Through study completion, assessed up to 3 years.
  The best overall response (BOR) is determined based on RECIST ver. 1.1, recorded from the start of protocol treatment. The determination of CR (Complete Response) and PR (Partial Response) shall be confirmed by the subsequent evaluation conducted at least 4 weeks after the criteria are first met.
Clinical Benefit Rate | Through study completion, assessed up to 3 years.
  The proportion of participants who achieved a best overall response of CR or PR according to RECIST version 1.1, or who maintained SD for 24 weeks or longer.
Clinical Benefit Duration | From enrollment to the end of treatment
  This is for participants who achieved the best overall response of CR or PR according to the RECIST version. 1.1, or who maintained SD for 24 weeks or longer, the period from the date of official registration (treatment initiation date) to the earliest date of determined disease progression, date of death due to any cause, or the end date of the clinical trial period.
Disease Control Rate | Through study completion, assessed up to 3 years.
  The proportion of participants who achieved the best overall response of CR or PR according to RECIST version. 1.1, or who maintained SD for 6 weeks or longer.
Progression-Free Survival | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  The period from the registration date as the starting point to the earlier of the date deemed as progression or the date of death due to any cause.
Overall Survival | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  The period from the registration date as the starting point until the date of death due to any cause. The last confirmed survival date is considered the cut-off point for surviving participants. For participants that become untraceable, the last date on which survival was confirmed before losing track is considered the cut-off point.
Adverse Event incidence | Through study completion, assessed up to 3 years
  Summarize and analyze the incidence and severity of adverse events. Evaluate the worst grade throughout all courses using CTCAE version. 5.0.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Jichi Medical University Hospital, Shimotsuke, Tochigi

IPD SHARING:
Plan to Share IPD: No